CLINICAL TRIAL: NCT06295666
Title: Gingival Crevicular Fluid(GCF) Bactericidal Permeability Protein (BPI) and Interleukin(IL)-1 Beta Levels and Relationship With Periodontal Disease
Brief Title: Gingival Crevicular Fluid (GCF) Bactericidal Permeability Protein (BPI) and Interleukin (IL)-1 Beta
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nezahat Arzu Kayar, Clinical Professor, Akdeniz University
Other Study IDs: 26.12.2018/901
Record Dates: First submitted 2024-01-02; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Periodontitis; Gingival Crevicular Fluid; Interleukin 1-beta; Bactericidal Permeability Protein
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gingival Crevicular Fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healty: Periodontal healty group
- Periodontitis: Periodontitis group

SUMMARY:
Objective: The aim of this study is to determine the amounts of BPI (Bactericidal permeability protein) and interleukin-1beta (IL-1β) in gingival fluid samples obtained from individuals with periodontally healthy and periodontal disease, to compare these amounts between study groups, and to evaluate their relationship with clinical parameters. In cases where clinical parameters increase, IL-1β amounts also increase significantly. The amount of IL-1β in individuals with periodontal disease is significantly higher compared to healthy individuals. There is positive correlation between BPI and clinical parameters. The amount of BPI in individuals with periodontal disease is significantly higher than in healthy individuals. More studies are needed to better understand the importance and therapeutic effect of BPI in periodontitis

DETAILED DESCRIPTION:
Systemically healthy and non-smoking participants were included in the study. The study groups included a total of 100 participants, 50 of whom were periodontally healthy (healthy group) and 50 with periodontal disease (periodontitis) group). The clinical parameters of plaque index (PI), gingival index (GI), and pocket depth (PD), clinical attachment level (CAL), and bleeding on probing (BOP) were measured.

The gingival fluid samples were taken in the direction of the paper strip and ELISA method was used for their analysis. A positive, statistically significant relationship was found between IL-1β levels and all clinical parameters (PI, GI, PD, CAL, BOP) (p<0,01). Likewise, there is a positive and significant relationship between BPI levels and clinical parameters (p<0,01).

There is a statistically significant positive correlation between GCF volume and clinical parameters PI (r: 0,722), GI (r: 0,740), PD (r: 0,742), CAL (r: 0,751) and BOP (r: 0.752) (p < 0.01). In the comparison between the groups, it is seen that both IL-1β and BPI levels were statistically significantly higher in the periodontitis group compared to the healthy group (p < 0,001).

ELIGIBILITY:
Inclusion Criteria:

1. For the periodontitis group, intraoral examination shows inflammation in the gums, supragingival and by observing the formation of subgingival tartar and microbial dental plaque and pockets, Diagnosis of periodontitis means that there is a vertical or detection of horizontal bone loss (Periodontitis group),
2. Failure to observe the presence of periodontal pockets, vertical and horizontal no bone destruction, bleeding score on full-mouth probing below 10 percent (Healthy group),
3. Agreeing to participate in the research and filling out and signing the voluntary consent form.

Exclusion Criteria:

1. Pregnant and lactating individuals,
2. Individuals who smoke,
3. Individuals with any systemic disease,
4. Individuals who have received periodontal treatment in the last 6 months,
5. Individuals who have used antibiotics in the last 6 months
6. Individuals in whom local factors that increase destruction such as fillings and crowns are observed in areas with periodontal pocket formation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who applied to Akdeniz University Faculty of Dentistry Department of Periodontology between 19/02/2019 and 25/11/2019 were included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Gingival Crevicular Fluid Bactericidal Permeability Increasing Protein levels in periodonitis | through study completion, an average of 1 year
  Protein levels that increase gingival crevicular fluid bactericidal permeability are expected to increase in the periodontitis group.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz Üniversitesi Diş Hekimliği Fakültesi, Antalya, Turkey (Türkiye)